CLINICAL TRIAL: NCT06451783
Title: The Clinical Efficacy of Shengyu Decoction Combined With Lijin Manipulation in the Treatment of Knee Osteoarthritis Was Observed Based on Three-dimensional Gait Analysis System
Brief Title: Shengyu Decoction and Lijin Manipulation for Knee OA: 3D Gait Analysis
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Principal Investigator, Liang Qiao, Clinical Professor, Xuhui Central Hospital, Shanghai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XuhuiCH202405
Record Dates: First submitted 2024-05-15; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Combined treatment group：Traditional Chinese medicine combined with manipulation treatment Control group：Oral control group medication
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined treatment group (Experimental): Traditional Chinese medicine combined with manipulation treatment：the Shengyu Decoction, which consists of the following herbs:
  * Shu Di Huang 20 grams
  * Bai Shao 15 grams
  * Dang Gui 15 grams
  * Chuan Xiong 8 grams
  * Ren Shen 20 grams
  * Huang Qi 18 grams One dose is taken per day, and a course of treatment consists of five weeks.
  Interventions: Other: Traditional Chinese medicine combined with manipulation treatment
- Control group (Active Comparator): Oral control group medication： Oral Celecoxib Capsules, 200mg per dose, once daily after lunch.
  Interventions: Drug: Celecoxib capsule

INTERVENTIONS:
Other: Traditional Chinese medicine combined with manipulation treatment — The specific procedure involves administering the Shengyu Decoction, which consists of the following herbs:
  * Shu Di Huang 20 grams
  * Bai Shao 15 grams
  * Dang Gui 15 grams
  * Chuan Xiong 8 grams
  * Ren Shen 20 grams
  * Huang Qi 18 grams One dose is taken per day, and a course of treatment consists of five weeks. Add manipulation of massage：
    * Press and grasp the affected limb three times；
      * Five-finger five-acupoint pressing method；
        * Point pressing on Zusanli (ST36) and Sanyinjiao (SP6)；
          * grasp the interior method to treat the calf three times；
            ⑤ Apply rolling technique around the knee joint；
            ⑥ Knead and straighten the standing tendon (the lateral muscle of the calf)；
            ⑦ Six-finger six-acupoint pressing method；
            ⑧ Push and pull the patella to flex and extend the knee joint；
            ⑨ Knee joint reunion and smooth dispersion method.
  Arms: Combined treatment group
Drug: Celecoxib capsule — Oral Celecoxib Capsules, 200mg per dose, once daily after lunch.
  Arms: Control group

SUMMARY:
Detailed Description Avoid duplicating information that will be entered or uploaded elsewhere in the record.

DETAILED DESCRIPTION:
This study aims to explore the efficacy of the Shengyu Decoction combined with manual therapy for the treatment of knee osteoarthritis (OA) using a clinical randomized controlled trial design. Additionally, based on three-dimensional gait analysis technology, the investigators will delve into the biomechanical mechanisms underlying the onset of knee OA and elucidate the mechanism of action of the Shengyu Decoction combined with manual therapy. This will further validate the clinical superiority of the Shengyu Decoction combined with manual therapy in the treatment of knee OA, providing strong support for reducing pain and improving knee function in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria of Western medicine: Knee pain for at least 1 month, X-ray showing osteophyte formation, age ≥50 years, morning stiffness ≤30 min, and bone fricative sound.
* TCM diagnostic criteria: Dull pain in the knee joint, flexion and extension limitations, pitching and side rotation unfavorability, slight activities slightly relieve pain, climate change aggravates symptoms, and repeated middle-aged and elderly patients, hidden onset, slow onset, slight local swelling of the knee joint, friction or clicking sound when moving, and severe cases may show muscle atrophy and joint deformity.
* Radiographs showing joint space narrowing, bone hyperplasia, subchondral osteosclerosis, and osteophyte formation.
* Patients who are between 45 and 85 years old.
* Patients who can understand and provide informed consent.
* Patients who are willing and able to undergo manual treatment for 1 course of treatment and cooperate with the doctor to complete the study.

Exclusion Criteria:

* Patients who do not meet the diagnostic criteria for knee osteoarthritis established by the rheumatology society.
* Severe knee pain with surgical indications (or X-ray grading standards reached level 4).
* Pregnant or planning to become pregnant.
* Patients who have participated in or are participating in other clinical trials within the last 3 months.
* Patients who have received or are receiving other treatment methods such as drugs that affect the evaluation of efficacy within the past 3 months.
* Patients with fractures, dislocation, skin damage, and severe infectious skin diseases within three weeks.
* Patients with severe primary diseases such as liver, kidney, hematopoietic system, endocrine system, cardiovascular and cerebrovascular, nervous system, tuberculosis, joint malformations, tumors, and psychiatric patients and postoperative patients.
* Patients who are unable to accurately evaluate the effectiveness and safety of treatment due to their medical condition.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The western Ontario and McMaster universities osteoarthritis index | up to 13 weeks
  The WOMAC consists of a series of questions that capture the patient's perception of pain, stiffness, and physical function over the past week. It is scored on a numerical scale, with higher scores indicating greater impairment. The index is often used in clinical trials and epidemiological studies to measure changes in osteoarthritis symptoms and to assess the effectiveness of treatments.

SECONDARY OUTCOMES:
Measurement of Gait Dynamics Parameters in Patients with Knee Osteoarthritis | up to 13 weeks
  Stride Length in meters
Measurement of Gait Dynamics Parameters in Patients with Knee Osteoarthritis | up to 13 weeks
  Walking Speed in meters per second
Gait Speed in meters per second | up to 13 weeks
  Gait Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Qiao Liang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No